CLINICAL TRIAL: NCT06644703
Title: Effect of Cryotherapy on Postoperative Pain in Vital Pulp Treatment of Molar Teeth With Symptomatic Irreversible Pulpitis: A Randomized Controlled Trial
Brief Title: Effect of Cryotherapy on Postoperative Pain in Vital Pulp Treatment of Molar Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Kübra Gürler, Cukurova University, Faculty of Dentistry, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 10.05.2025/144
Record Dates: First submitted 2024-10-01; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Pulpitis - Irreversible
Keywords: Cryotherapy; Vital pulp therapy; Irreversibl pulpitis; Postoperative pain; Total pulpotomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy group (Experimental): After the coronal pulp tissue was completely removed up to the root canal orifice with a high-speed sterile diamond bur under water cooling, hemostasis was achieved within 8 minutes using a cotton pellet moistened with 1% NaOCl. The pulpotomy area was irrigated with 2 °C saline solution for 5 minutes. Then, the pulp chamber was covered with 2-3 mm thick Bio MTA+ (Cerkamed Company, Poland) and composite restoration of the teeth (Clearfil Majesty Posterior, Kuraray Medical Inc, Tokyo, Japan) was completed in the same visit.
  Interventions: Other: Cryotherapy
- Control group (No Intervention): After the coronal pulp tissue was completely removed up to the root canal orifice with a high-speed sterile diamond bur under water cooling, hemostasis was achieved within 8 minutes using a cotton pellet moistened with 1% NaOCl. Then, the pulp chamber was covered with 2-3 mm thick Bio MTA+ (Cerkamed Company, Poland) and composite restoration of the teeth (Clearfil Majesty Posterior, Kuraray Medical Inc, Tokyo, Japan) was completed in the same visit.

INTERVENTIONS:
Other: Cryotherapy — The pulpotomy area was irrigated with 2 °C saline solution for 5 minutes in cryotherapy group.
  Arms: Cryotherapy group

SUMMARY:
The goal of this clinical trial was to evaluate the effect of cryotherapy with salin solution on the intensity of postoperative pain after total pulpotomy procedures in molar teeth with symptomatic irreversible pulpitis. The main question it aims to answer is:

- Does controlled irrigation with cold saline in total pulpotomy reduce the severity of postoperative pain? In the cryotherapy group, unlike the control group, after hemostasis was achieved, the coronal pulp cavity was irrigated with 2 °C saline solution for 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

Teeth with

* moderate or severe pain
* diagnosed with symptomatic irreversible pulpitis
* no tenderness to percussion and palpation
* positive response to cold test and electric pulp test
* no signs of periapical pathology

Exclusion Criteria:

Teeth which

* could not be restored or required post-core
* had periapical lesions,
* had poor periodontal status (pocket depth> 4 mm),
* had negative responses to pulp sensitivity tests,
* had no pulp exposure after caries removing Patients who
* had no preoperative pain or had mild preoperative pain
* had bleeding disorders
* had systemic diseases such as immunosuppressive disease or diabetes

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | up to 72 hours
  The visual analog scale for pain is a straight line with one end meaning no pain (0) and the other end meaning the worst pain (10) imaginable. A patient marks a point on the line that matches the amount of pain he or she feels. It may be used to help choose the right dose of pain medicine. Also called VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Hamdi Oğuz Yoldaş, DDS PHD, Study Director — Cukurova University
Locations (1):
- Çukurova Üniversitesi Diş Hekimliği Fakültesi, Gültepe, Sarıçam/Adana/Türkiye, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akhil VS, Kumar V, Aravind A, Sharma R, Sharma S, Chawla A, Upadhyay AD, Logani A. Novel cryotherapy technique for pulpotomy in mature permanent teeth with symptomatic irreversible pulpitis- a randomized controlled trial. Clin Oral Investig. 2024 Apr 26;28(5):275. doi: 10.1007/s00784-024-05661-y. PMID 38668793
- [Background] Keskin C, Ozdemir O, Uzun I, Guler B. Effect of intracanal cryotherapy on pain after single-visit root canal treatment. Aust Endod J. 2017 Aug;43(2):83-88. doi: 10.1111/aej.12175. Epub 2016 Oct 4. PMID 27699913